CLINICAL TRIAL: NCT01874717
Title: Conscious Sedation With Midazolam in Dentally Anxious Patients: Effect of the Administration Route (Oral Versus Intravenous Administration)
Brief Title: Midazolam Sedation in Dentally Anxious Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CHU-0155
Record Dates: First submitted 2013-05-28; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Dental Anxiety
Keywords: Conscious sedation; Dental anxiety; Oral midazolam; Intravenous midazolam; Behaviour
MeSH Terms: conditions — Behavior | interventions — Conscious Sedation; Dental Care; Midazolam

ARMS (2):
- oral midazolam (Experimental): oral administration of midazolam : the dose administered is twice the individual dose determined in session 1.
  Interventions: Other: Conscious sedation for dental care; Drug: midazolam
- intravenous midazolam (Other): intravenous administration of midazolam at the individual dose determined in session 1
  Interventions: Other: Conscious sedation for dental care; Drug: midazolam

INTERVENTIONS:
Other: Conscious sedation for dental care
Drug: midazolam

SUMMARY:
Use lay language.

To compare patient level of cooperation during dental care under conscious sedation with midazolam according to the administration route

DETAILED DESCRIPTION:
The progress of the study is described below:

Session 1: intravenous administration of midazolam. Establishment of the individual dose.

Randomisation.

Session 2 :

Group A : oral administration of midazolam : the dose administered is twice the individual dose determined in session 1.

Group B : intravenous administration of midazolam at the individual dose determined in session 1.

Session 3 : reversal of the procedures :

Group A : intravenous administration of midazolam at the individual dose determined in session 1.

Group B : oral administration of midazolam : the dose administered is twice the individual dose determined in session 1.

ELIGIBILITY:
Inclusion Criteria:

* - Patient between 8 and 60 years, regardless of gender
* Patient in the American Society of Anesthesiologists (ASA) category I ou II.
* Patient in need of multiple dental care, referred to the Unit of Special Care Dentistry for cooperation difficulties
* Patients directed to conscious sedation under midazolam because they cannot be approached for more than a very brief examination, or following failure to treat under inhalation sedation (50% N2O/O2), or following poor cooperation during treatment under inhalation sedation (poor cooperation is defined as a score of 3 or more on the French modified version of the Venham scale), or following good cooperation during short and simple treatment under inhalation sedation but in need of more complex rehabilitation.
* Written consent signed by the patient or his legal guardian
* Patient accompanied by an accountable person

Exclusion Criteria:

* - Patient below 8 years or over 60 years-old
* Patient in the American Society of Anesthesiologists (ASA) category III or more
* Patient having accepted dental treatment without premedication or sedation, and without declaring dental anxiety, during the month prior to the appointment
* Patient having received an anxiolytic premedication in the 24 hours preceding the dental care session
* Patient already treated under midazolam sedation less than a week ago
* Any medical contraindication to the use of midazolam

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 131 (Actual)
Dates: Start 2005-06; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Patient level of cooperation which is assessed using the French modified version of Venham scale | At the first contact with the dentist (at day 1)
  This scale offers a good description of behaviour and anxiety in one score (from0 to 5)
Patient level of cooperation which is assessed using the French modified version of Venham scale | During venous cannulation (at day 1)
  This scale offers a good description of behaviour and anxiety in one score (from 0 to 5)
Patient level of cooperation which is assessed using the French modified version of Venham scale | During the first injection of local anaesthesia (at day 1)
  This scale offers a good description of behaviour and anxiety in one score (from0 to 5)
Patient level of cooperation which is assessed using the French modified version of Venham scale | During the first dental care procedure (at day 1)
  This scale offers a good description of behaviour and anxiety in one score (from0 to 5)

SECONDARY OUTCOMES:
The level of patient stress which is assessed using the French modified version of Venham scale | at T1 (first contact)
  This scale offers a good description of behaviour and anxiety in one score (from0 to 5)
The level of patient stress which is assessed using the French modified version of Venham scale | at T8 (end of dental treatment)
  This scale offers a good description of behaviour and anxiety in one score (from0 to 5)
Satisfaction level of the patient which is assessed using the French modified version of Venham scale | 48 hours after dental care (T14).
  This scale offers a good description of behaviour and anxiety in one score (from 0 to 5)
Satisfaction level of the accompanying person which is assessed using the French modified version of Venham scale | 48 hours after dental care (T14).
  This scale offers a good description of behaviour and anxiety in one score (from 0 to 5)
Satisfaction level of the operator which is assessed using the French modified version of Venham scale | 48 hours after dental care (T14).
  This scale offers a good description of behaviour and anxiety in one score (from 0 to 5)

CONTACTS AND LOCATIONS:
Overall Officials: Valérie COLLADO, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Collado V, Faulks D, Nicolas E, Hennequin M. Conscious sedation procedures using intravenous midazolam for dental care in patients with different cognitive profiles: a prospective study of effectiveness and safety. PLoS One. 2013 Aug 5;8(8):e71240. doi: 10.1371/journal.pone.0071240. Print 2013. PMID 23940729